CLINICAL TRIAL: NCT06916546
Title: Yttrium-90 Selective Internal Radiation Therapy (SIRT) Combined With Lenvatinib and PD-(L)1 Inhibitors Versus Transarterial Chemoembolization (TACE) Combined With Lenvatinib and PD-(L)1 Inhibitors for Intermediate-Advanced Hepatocellular Carcinoma: A Multicenter Retrospective Study
Brief Title: SIRT or TACE Plus Lenvatinib and PD-(L)1 Inhibitor in High Burden HCC
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Jinshazhou Hospital of Guangzhou University of Chinese Medicine (Unknown); First Affiliated Hospital of Army Military Medical University (Unknown); Hainan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MIIR-25-retro
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: hepatocellular carcinoma; selective internal radiation therapy; transarterial chemoembolization; lenvatinib; PD-(L)1 Inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SIRT-L-P: Patients were treated with SIRT-L-P
  Interventions: Combination Product: SIRT-L-P
- TACE-L-P: Patients were treated with TACE-L-P
  Interventions: Combination Product: TACE-L-P

INTERVENTIONS:
Combination Product: SIRT-L-P — Patients received 1-2 session of SIRT. Lenvatinib and PD-(L)1 inhibitor was initiated within 7 days after the first SIRT and continued until unacceptable toxicity, disease progression, initiation of new therapy, or loss to follow-up.
  Groups: SIRT-L-P
Combination Product: TACE-L-P — Patients received TACE. TACE was repeated for viable tumors demonstrated by follow-up imaging in patients without worsening liver function or contraindications (on-demand TACE). Lenvatinib and PD-(L)1 inhibitor was initiated within 7 days after the first SIRT and continued until unacceptable toxicity, disease progression, initiation of new therapy, or loss to follow-up.
  Groups: TACE-L-P

SUMMARY:
This multicenter retrospective study evaluated the efficacy and safety of selective internal radiation therapy (SIRT) combined with lenvatinib and PD-(L)1 inhibitors (SIRT-L-P) versus transarterial chemoembolization (TACE) combined with lenvatinib and PD-(L)1 inhibitors (TACE-L-P) in patients with HCC beyond up-to-seven criteria or with portal vein tumor thrombus (PVTT). Tumor response, progression-free survival (PFS), overall survival (OS), and adverse events (AEs) were compared between the two groups.

DETAILED DESCRIPTION:
Consecutive patients with HCC beyond up-to-seven criteria or with PVTT treated with SIRT-L-P or TACE-L-P from June 2022 to October 2024 were screened. Tumor response was evaluated according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) and Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1). Clinical outcomes, including tumor response, PFS, OS, and AEs were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* histologically or clinically confirmed diagnosis of HCC at BCLC stage B or C (extrahepatic metastases were allowed)
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1
* Child-Pugh class A or B7
* unresectable HCC with intrahepatic tumor beyond up-to-seven criteria and/or with PVTT.

Exclusion Criteria:

* receipt of other loco-regional therapies, including hepatic arterial infusion chemotherapy, external radiation therapy, or radioactive seed implantation
* Prior systemic therapy
* History of other malignancies
* incomplete medical records

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate-advanced HCC beyond up-to-seven criteria and/or with PVTT.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 32 months
  The time from the first SIRT or TACE procedure until the date that progressive disease according to mRECIST or death was confirmed.

SECONDARY OUTCOMES:
Objective response rate (ORR) | 32 months
  the percentage of patients with complete or partial response according to mRECIST and RECIST 1.1
Overall survival | 32 months
  the time from the first SIRT or TACE until the date of all-cause mortality
Disease control rate (DCR) | 32 months
  the percentage of patients with complete, partial response, or stable disease according to mRECIST and RECIST 1.1

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No